CLINICAL TRIAL: NCT06984289
Title: Role of Radiomics Applied to Ultrasound in Patients With Locally Advanced Cervical Cancer: a Retrospective Multicenter Study
Brief Title: US Radiomics in Advanced Cervical Cancer
Acronym: RU-LACC
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7443
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Uterine Cervical Neoplasms; Locally Advanced Cervical Cancer; Radiomics; Ultrasound Imaging; Machine Learning; Chemoradiotherapy
Keywords: Locally Advanced Cervical Cancer; Cervical Cancer; Uterine Cervical Neoplasms; Radiomics; Ultrasound; Ultrasound Imaging; Machine Learning; Gynecologic Oncology
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Responder Group: Patients with locally advanced cervical cancer who responded to primary treatment (either exclusive chemoradiotherapy or neoadjuvant chemoradiotherapy followed by radical surgery), as determined by clinical and/or histological assessment.
  Interventions: Other: Radiomic Analysis of Ultrasound Images
- Non-Responder Group: Patients with locally advanced cervical cancer who did not respond to primary treatment (either exclusive chemoradiotherapy or neoadjuvant chemoradiotherapy followed by radical surgery), based on residual disease findings or lack of clinical response.
  Interventions: Other: Radiomic Analysis of Ultrasound Images

INTERVENTIONS:
Other: Radiomic Analysis of Ultrasound Images — Quantitative analysis of pre-treatment ultrasound images of the primary cervical tumor to extract radiomic features. These features will be used to develop and validate machine learning models for predicting treatment response and disease relapse in patients with locally advanced cervical cancer (LACC).
  Other Names: Radiomics, Ultrasound-based Radiomics, Radiomic Feature Extraction

SUMMARY:
This is a retrospective, multicenter observational study aimed at evaluating the role of ultrasound-based radiomics in patients with locally advanced cervical cancer (LACC). The study will analyze pre-treatment ultrasound images to identify radiomic features that may predict treatment response and disease recurrence.

A total of 220 patients treated with exclusive chemoradiotherapy or neoadjuvant chemoradiotherapy followed by radical surgery between 2011 and 2024 will be included. Using clinical and imaging data, machine learning models will be developed to distinguish between responders and non-responders, and to identify patients at higher risk of relapse.

The goal is to improve personalized care in LACC by integrating radiomic analysis into treatment planning and follow-up strategies.

ELIGIBILITY:
Inclusion Criteria:

Female patients aged ≥18 years

Histologically confirmed diagnosis of locally advanced cervical cancer (FIGO 2018 stage IB3-IVA, excluding IIA1)

Histologic subtypes: squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma

Underwent transvaginal or transrectal ultrasound prior to treatment

At least one pre-treatment DICOM ultrasound image of the primary tumor available

Treated with either exclusive chemoradiotherapy or neoadjuvant chemoradiotherapy followed by radical surgery

Completed at least 12 months of follow-up after primary treatment

Signed informed consent (or equivalent declaration)

Exclusion Criteria:

Age <18 years

Only printed ultrasound images available

Ultrasound images with poor tumor visualization or with text/markers obscuring the tumor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced cervical cancer (FIGO 2018 IB3-IVA, excluding IIA1), treated between 2011 and 2024, from multiple Italian centers. All participants underwent ultrasound before treatment and have available DICOM images for radiomic analysis.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2025-03-25 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-14 (Actual)

PRIMARY OUTCOMES:
Performance of ultrasound-based radiomic models in predicting treatment response in patients with locally advanced cervical cancer. | Up to 12 months after primary treatment.
  Evaluation of the diagnostic accuracy (AUC, sensitivity, specificity, F1-score) of radiomic models based on pre-treatment ultrasound images in distinguishing responder vs. non-responder patients to primary treatment (exclusive chemoradiotherapy or neoadjuvant chemoradiotherapy followed by radical surgery). Models will be developed and validated using retrospective data.

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Culcasi, Study Chair — Fondazione Policlinico Universitario Agostino Gemelli
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No